CLINICAL TRIAL: NCT02848625
Title: Yoga Effect on Quality of Life Study Among Patients with Idiopathic Pulmonary Fibrosis
Acronym: YES-IPF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ganesh Raghu, Co-Principal Investigator (Ganesh Raghu, MD is Principal Investigator), University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 51411-A
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Yoga; Quality of life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Patients randomized to 12 weeks of twice weekly yoga sessions. The yoga exercises have been designed specifically for patients with IPF. Yoga sessions were virtual in the setting of the COVID Pandemic
  Interventions: Other: Yoga
- Group B (No Intervention): Patients who are not randomized to yoga sessions will continue with their usual care and usual activities

INTERVENTIONS:
Other: Yoga — Yoga and breathing exercises designed for patients with IPF. Sessions will be two times per week for 12 weeks
  Arms: Group A

SUMMARY:
This study will evaluate whether regular yoga exercises designed specifically for patients with Idiopathic Pulmonary Fibrosis is associated with any change in quality of life. Half of the participants will be randomized to yoga, half to usual care. Yoga was conducted live, virtually, in the setting of the COVID Pandemic.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis (IPF) is a chronic progressive fibrotic (scarring) disease of the lung of unknown cause. Approximately 100,000 Americans will die from IPF this year. There is no cure for IPF other than lung transplantation, which only 1% of patients will receive. Recently, 2 drugs were approved by the FDA to slow the rate of decline in lung function among patients with IPF. These drugs do not decrease symptoms or improve quality of life.

Symptoms of IPF include shortness of breath, cough, and fatigue, all of which may also adversely affect quality of life. Yoga is a practice of exercises, including breathing exercises, that has been shown to be relatively safe and to improve quality of life in some patients with other advanced lung diseases. We hypothesize that regular yoga and breathing exercises, specifically designed for patients with Idiopathic Pulmonary Fibrosis, over a period of 12 weeks will lead to improved quality of life as measured by several different quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria: Adults 18 years of age or older. We will include all consecutive consenting patients with IPF who are able to provide informed consent and are seen and followed at the Center for Interstitial Lung Disease at the University of Washington Medical Center.

Exclusion Criteria: Subjects with comorbid diseases that would prohibit them from taking part in yoga will be excluded at the discretion of the clinical-investigators. Such comorbid diseases would include paralysis, musculoskeletal discomfort that would interfere with participation or broken limbs. Since we are interested in the effect of yoga among subjects with IPF, we will exclude subjects who have previously received lung transplantation. To assess the effect "new" or "initial" participation in a yoga program with breathing exercises on quality of life, subjects who are regularly participating in yoga (outside of the study) will be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 12 weeks

SECONDARY OUTCOMES:
change in forced vital capacity | 12 weeks
change in 6 minute walk distance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Raghu, MD, Principal Investigator — University of Washington, Center for Interstitial Lung Diseases; Bridget F Collins, MD, Principal Investigator — University of Washington, Center for Interstitial Lung Diseases
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No